CLINICAL TRIAL: NCT02244918
Title: Informing Tobacco Treatment Guidelines for African American Non-Daily Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001602; AD-1310-08709 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Active Comparator): Participants will go to smoking cessation counseling over 12 weeks. They will be asked to participated in 5 total counseling sessions.
  Interventions: Behavioral: Smoking Cessation Counseling
- Counseling Plus NRT (Experimental): Participants will go to smoking cessation counseling over 12 weeks. They will be asked to participated in 5 total counseling sessions. In addition to counseling, participants in this group will also take 12 weeks of a nicotine replacement therapy(NRT) (like the patch, gum or lozenge) of their choice.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — Participant has choice of from over-the-counter nicotine patch, nicotine gum or lozenge.
  Arms: Counseling Plus NRT
Behavioral: Smoking Cessation Counseling

SUMMARY:
The researchers are testing if counseling alone or counseling plus over-the-counter nicotine replacement therapies (NRT), like the patch,gum, or lozenge, helps African American non-daily smokers quit smoking.

DETAILED DESCRIPTION:
Non-daily smokers represent a growing number of racial/ethnic minority smokers. 1 out of 4 African Americans are non-daily smokers. African Americans seem to have a harder time quitting and have greater medical problems related to smoking even at lighter usage rates compared to Whites.

Current tobacco treatment guidelines target daily smokers. There are no guidelines for non-daily smokers. This study will allow the researchers to explore treatment options for African American non-daily smokers and find out if some treatments work better than others.

Participation in this study will last about 6 months. Over this course of time, participants will be asked to visit the study location 3 times and will talk with a member of the study team on the phone 4 times.

ELIGIBILITY:
Inclusion Criteria:

* African American adults who are interested in quitting and whose smoking patterns meet criteria for non-daily smoking as determined by eligibility screening

Exclusion Criteria:

* Contraindications to behavioral counseling, nicotine gum, patch, or lozenge and unable to complete study procedures as determined by eligibility screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11-01 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Nollen, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Swope Health Central, Kansas City, Missouri

REFERENCES:
- [Derived] Nollen NL, Cox LS, Mayo MS, Ellerbeck EF, Madhusudhana S, Ahluwalia JS. A randomized clinical trial of counseling and nicotine replacement therapy for treatment of African American non-daily smokers: Design, accrual, and baseline characteristics. Contemp Clin Trials. 2018 Jul;70:72-82. doi: 10.1016/j.cct.2018.05.011. Epub 2018 May 19. PMID 29787858

RESULTS

PARTICIPANT FLOW:
Groups:
- Counseling Plus Nicotine Replacement Therapy: Participants will attend 5 smoking cessation counseling sessions over 12 weeks.In addition to counseling, participants in this group will also take 12 weeks of a nicotine replacement therapy (like the patch, gum or lozenge) of their choice.
  Nicotine Replacement Therapy: Participant has choice of from over-the-counter nicotine patch, nicotine gum or lozenge.
- Counseling: Participants will attend 5 smoking cessation counseling sessions over 12 weeks.
Period: Overall Study
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Started | 185 | 93
Week 12 (End of Treatment) | 160 | 83
Completed | 185 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Counseling Plus Nicotine Replacement Therapy: Participants will attend 5 smoking cessation counseling sessions over 12 weeks. In addition to counseling, participants in this group will also take 12 weeks of a nicotine replacement therapy (like the patch, gum or lozenge) of their choice.
  Nicotine Replacement Therapy: Participant has choice of from over-the-counter nicotine patch, nicotine gum or lozenge.
- Total: Total of all reporting groups
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling | Total
Number analyzed (Participants) | 185 | 93 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (1.6) | 49 (11.8) | 48.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 47 | 141
  Male | 91 | 46 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American, Non-Hispanic | 185 | 93 | 278
Region of Enrollment [Number; unit: participants]
  United States | 185 | 93 | 278
Cohabitation Status, Married or living with a partner [Count of Participants; unit: Participants] | 48 | 17 | 65
Employed Full-time [Count of Participants; unit: Participants] | 45 | 29 | 74
Education level of less than High School graduate [Count of Participants; unit: Participants] | 27 | 13 | 40
Has health insurance [Count of Participants; unit: Participants] | 146 | 67 | 213
< or = 100% Poverty Level [Count of Participants; unit: Participants] | 79 | 38 | 117
Own a Home [Count of Participants; unit: Participants] | 25 | 7 | 32
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (8.7) | 31.7 (9.8) | 31.5 (9.1)
Days smoked cigarettes in the last 30 [Mean (Standard Deviation); unit: days] | 23.2 (8.0) | 22.8 (8.0) | 23.1 (8.0)
Number of cigarettes used on days smoked [Mean (Standard Deviation); unit: cigarettes] | 4.8 (3.6) | 4.4 (3.2) | 4.7 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Biochemically confirmed 30-day point prevalence abstinence at Week 12 using urine anabasine and anatabine, with the recommended cut-off of 2 ng/ml to differentiate smokers from non-smokers.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
Participants | 21 | 8

2. Secondary Outcome: Smoking Abstinence
Description: Biochemically confirmed 30-day point prevalence abstinence at Week 26 using urinary cotinine, with the recommended cut-off of 50 ng/ml to differentiate smokers from non-smokers.
Time Frame: Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
Participants | 13 | 6

3. Secondary Outcome: Concentration of Urinary Cotinine
Description: Measured by urinary cotinine, a biochemical marker of nicotine intake, sampled from participants at weeks 0 and 26.
Time Frame: Weeks 0, 26
Population: Number analyzed at the week 26 follow-up time point reflects the number of participants who returned for this visit.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
ng/ml
  Baseline Nicotine Exposure | 1538.3 (1622.0) | 1905.3 (1695.3)
  Week 26 Nicotine Exposure: number analyzed (Participants) | 128 | 74
  Week 26 Nicotine Exposure | 1513.2 (1779.0) | 1649.3 (1443.9)

4. Secondary Outcome: Urinary Concentration of NNAL (4-(Methyl Nitrosamine)-1-(3-pyridyl)-1-butanol)
Description: Measured by a change in NNAL (4-(methyl nitrosamine)-1-(3-pyridyl)-1-butanol),a biochemical marker of tobacco-specific carcinogen exposure. Levels assessed by urine sample from each participant and Weeks 0 and 12.
Time Frame: Weeks 0, 12
Population: The number of participants analyzed at follow-up time-points reflects only those who returned at that point.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
pg/ml
  Baseline Carcinogen Exposure | 100.9 (121.0) | 97.1 (97.8)
  Week 12 Carcinogen Exposure: number analyzed (Participants) | 158 | 83
  Week 12 Carcinogen Exposure | 47.6 (55.2) | 49.3 (47.3)

5. Secondary Outcome: Total Days Abstinent
Description: Number of days abstinent from baseline through week 26.
Time Frame: Week 0-26
Population: The number of participants analyzed at follow-up time-points reflects only those who returned at that point.
Measure: Mean (Standard Deviation); unit: days abstinent in the past 30 days
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
days abstinent in the past 30 days
  Baseline days abstinent from all tobacco | 10.3 (6.4) | 10.4 (6.4)
  Week 4 days abstinent from all tobacco: number analyzed (Participants) | 162 | 81
  Week 4 days abstinent from all tobacco | 17.4 (9.0) | 12.8 (9.2)
  Week 8 days abstinent from all tobacco: number analyzed (Participants) | 154 | 81
  Week 8 days abstinent from all tobacco | 20.8 (9.0) | 19.8 (10.7)
  Week 12 days abstinent from all tobacco: number analyzed (Participants) | 160 | 83
  Week 12 days abstinent from all tobacco | 19.8 (10.7) | 14.8 (11.1)
  Week 26 days abstinent from all tobacco: number analyzed (Participants) | 132 | 75
  Week 26 days abstinent from all tobacco | 19.2 (11.2) | 15.1 (11.2)

6. Secondary Outcome: Cigarettes Used
Description: Cigarettes used in the past 30 days from baseline through week 26
Time Frame: Weeks 0-26
Population: The number of participants analyzed at follow-up time-points reflects only those who returned at that point.
Measure: Mean (Standard Deviation); unit: Cigarettes used in the past 30 days
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
Number analyzed (Participants) | 185 | 93
Cigarettes used in the past 30 days
  Baseline | 100.4 (102.1) | 85.8 (72.6)
  Week 4: number analyzed (Participants) | 162 | 81
  Week 4 | 43.2 (58.5) | 57.9 (51.8)
  Week 8: number analyzed (Participants) | 154 | 81
  Week 8 | 30.9 (52.3) | 53.3 (64.3)
  Week 12: number analyzed (Participants) | 160 | 83
  Week 12 | 37.1 (69.4) | 49.0 (56.6)
  Week 26: number analyzed (Participants) | 132 | 75
  Week 26 | 46.9 (81.0) | 48.7 (57.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 12 weeks.
Description: At each assessment point, participants were asked to report any new or worsening symptoms.
Arm/Group | Counseling Plus Nicotine Replacement Therapy | Counseling
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/93
Other Adverse Events (participants affected / at risk) | 161/185 | 83/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Counseling Plus Nicotine Replacement Therapy (N=185) | Counseling (N=93)
Breathing Problems (Respiratory, thoracic and mediastinal disorders) | 59 | 28
Blisters in the mouth, increased saliva, or other problems with the mouth, tooth or jaw (Gastrointestinal disorders) | 59 | 20
Bowel changes like constipation or diarrhea (Gastrointestinal disorders) | 70 | 36
Changes in taste (Gastrointestinal disorders) | 104 | 45
Cold Sweats or increased sweating (Endocrine disorders) | 72 | 34
Difficulty concentrating or confusion.mental weakness (Psychiatric disorders) | 63 | 34
Disturbed hearing or vision (Ear and labyrinth disorders) | 37 | 24
Dizziness (Ear and labyrinth disorders) | 51 | 21
Headache (General disorders) | 87 | 44
Heartburn, indigestion, hiccups or burping (Gastrointestinal disorders) | 88 | 43
Irregular or fast heart beat (Cardiac disorders) | 40 | 20
Irritability (General disorders) | 105 | 63
Nausea or vomiting (Gastrointestinal disorders) | 53 | 17
Nervous, restless, anxious (Nervous system disorders) | 103 | 56
Redness/swelling/rash/irritation on the skin (Skin and subcutaneous tissue disorders) | 36 | 6
Sleeping Problems (General disorders) | 98 | 56
Sore throat (Gastrointestinal disorders) | 43 | 19
Stomach cramps or pains (Gastrointestinal disorders) | 40 | 0
Tiredness/fatigue (General disorders) | 109 | 67

LIMITATIONS AND CAVEATS:
Findings may not generalize to non-daily smokers of other racial/ethnic groups. Low rates of cessation overall limited the potential for analyses of differential effects in sub-populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02244918/Prot_SAP_000.pdf